CLINICAL TRIAL: NCT00336453
Title: Evaluation of the Safety, Reactogenicity and Immunogenicity of FluBlok Trivalent Recombinant Baculovirus-Expressed Hemagglutinin Influenza Vaccine Administered Intramuscularly to Healthy Children Aged 6 To 59 Months
Brief Title: Immunogenicity and Safety of FluBlok Trivalent Recombinant Hemagglutinin Influenza Vaccine in Healthy Pediatrics
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Protein Sciences Corporation (Industry)
Responsible Party: Manon Cox, Chief Operating Officer, Protein Sciences Corporation
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: PSC02
Record Dates: First submitted 2006-06-12; First posted 2006-06-13 (Estimated); Last update posted 2009-12-17 (Estimated); Status verified 2009-12

CONDITIONS: Influenza
Keywords: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines; FluBlok

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- FluBlok-22.5 μg, 6-35 months old (Experimental): 6-35 months old, FluBlok-22.5 μg of each recombinant hemagglutinin antigen: 2006-2007 formulation containing A/New Caledonia/20/99 (H1N1), A/Wisconsin/67/05 (H3N2), and B/Ohio/01/05 like viruses
  Interventions: Biological: Influenza Vaccination
- FluBlok-45 μg, 6-35 months old (Experimental): 6-35 months old, FluBlok-45 μg of each recombinant hemagglutinin antigen: 2006-2007 formulation containing A/New Caledonia/20/99 (H1N1), A/Wisconsin/67/05 (H3N2), and B/Ohio/01/05 like viruses
  Interventions: Biological: Influenza Vaccination
- TIV-7.5 μg, 6-35 months old (Active Comparator): 6-35 months old, 2006-2007 formulation of Fluzone, (sanofi-pasteur, Swiftwater, PA)-7.5 μg of each hemagglutinin antigen: A/New Caledonia/20/99 (H1N1), A/Wisconsin/67/05 (H3N2), and B/Malaysia/2506/2004 like viruses
  Interventions: Biological: Influenza Vaccination
- TIV-15 μg, 36-59 months old (Active Comparator): 36-59 months old, 2006-2007 formulation of Fluzone (sanofi-pasteur, Swiftwater, PA)-15 μg of each hemagglutinin antigen: A/New Caledonia/20/99 (H1N1), A/Wisconsin/67/05 (H3N2), and B/Malaysia/2506/2004 like viruses
  Interventions: Biological: Influenza Vaccination
- FluBlok-45 μg, 36-59 months old (Experimental): 36-59 months old, FluBlok-45 μg of each recombinant hemagglutinin antigen: 2006-2007 formulation containing A/New Caledonia/20/99 (H1N1), A/Wisconsin/67/05 (H3N2), and B/Ohio/01/05 like viruses
  Interventions: Biological: Influenza Vaccination

INTERVENTIONS:
Biological: Influenza Vaccination — 0.5mL dose for intramuscular injection
  Other Names: FluBlok; Fluzone; rHA; rHA0; recombinant hemagglutinin; TIV
  Arms: FluBlok-45 μg, 36-59 months old; FluBlok-45 μg, 6-35 months old; TIV-15 μg, 36-59 months old
Biological: Influenza Vaccination — 0.25mL dose for intramuscular injection
  Other Names: FluBlok; Fluzone; rHA; rHA0; recombinant hemagglutinin; TIV
  Arms: FluBlok-22.5 μg, 6-35 months old; TIV-7.5 μg, 6-35 months old

SUMMARY:
The purpose of this study was to evaluate dose-related safety, reactogenicity and immunogenicity of FluBlok trivalent recombinant baculovirus-expressed hemagglutinin influenza vaccine, administered to healthy children aged 6 to 59 months.

DETAILED DESCRIPTION:
Influenza has been identified as a major health problem in young children. Influenza related hospitalizations are very high in children less than 24 months of age and children age 24-59 months have a high rate of medical care utilization due to influenza. Recently, it has been noted that there are deaths attributable to influenza even in previously healthy children. Recent CDC recommendations reflect this growing awareness of the impact of influenza in children and state that virtually all children less than 18 years of age should receive annual influenza vaccination.

Currently available licensed trivalent influenza vaccines (TIVs) are prepared from viruses that are grown in embryonated hens' eggs. Alternative substrates for vaccine production are desirable in order to reduce the vulnerability of and to expand influenza vaccine supply. Recombinant DNA techniques allow for expression of the influenza hemagglutinin (rHA) by baculovirus vectors in insect cell cultures. Advantages of this technique include speed of production, absence of egg protein, and a highly purified product.

ELIGIBILITY:
Inclusion Criteria:

1. The subject was:

   1. aged 6-59 months old (inclusive) at enrollment.
   2. in good health (and not on any chronic medications), as determined by medical history and a history directed targeted physical examination.
   3. naïve for previous influenza vaccination prior to study enrollment.
2. Parents or guardians must:

   1. be able to understand and comply with planned study procedures and be available for all study visits.
   2. provide written consent prior to initiation of any study procedures, and subject may provide written assent as appropriate.

Exclusion Criteria:

1. a known allergy to eggs or other components of the vaccine or sensitivity or allergy to latex.
2. a history of severe asthma or more than three previous wheezing episodes.
3. be undergoing immunosuppression as a result of an underlying illness or treatment.
4. an active neoplastic disease or a history of any hematologic malignancy.
5. be using oral or parenteral steroids, inhaled steroids or other immunosuppressive or cytotoxic drugs. Note: Subjects on nasal or topical steroids will be allowed to enroll in this study.
6. a history of receiving influenza vaccine or plans during the study to receive influenza vaccine outside the study.
7. a history of receiving immunoglobulin or other blood product within the 3 months prior to enrollment in this study.
8. received any other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrollment in this study.
9. have an acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe or would interfere with the evaluation of responses (these conditions include, but are not limited to: known chronic liver disease, significant renal disease, unstable or progressive neurological disorders, diabetes mellitus, and transplant recipients).
10. a history of severe reactions following immunization.
11. an acute illness, including an axillary temperature greater than 100.0*F, within 3 days prior to vaccination.
12. received an experimental vaccine or medication within 1 month prior to enrollment in this study, or expect to receive an experimental vaccine, medication, or blood product during the 6-month study period.
13. any condition that would, in the opinion of the investigator, place them at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.
14. a history of Guillain-Barré syndrome.
15. be participating concurrently in another clinical trial (either in active phase or in follow-up phase).

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 156 (Actual)
Dates: Start 2006-10; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of safety and reactogenicity of FluBlok and TIV in healthy children aged 6-59 months | influenza season

SECONDARY OUTCOMES:
To compare the immunogenicity after each dose of two different formulations of FluBlok to TIV in healthy children aged 6-35 months and one formulation of FluBlok to TIV in healthy children aged 36-59 months. | Day 0, 28, 56

CONTACTS AND LOCATIONS:
Overall Officials: James C King, MD, Principal Investigator — University of Maryland
Locations (3):
- United States (3):
  - Kentucky pediatric /Adult Research, Bardstown, Kentucky
  - Saint Louis University, St Louis, Missouri
  - Primary Physicians Research, Pittsburgh, Pennsylvania

REFERENCES:
- [Result] King JC Jr, Cox MM, Reisinger K, Hedrick J, Graham I, Patriarca P. Evaluation of the safety, reactogenicity and immunogenicity of FluBlok trivalent recombinant baculovirus-expressed hemagglutinin influenza vaccine administered intramuscularly to healthy children aged 6-59 months. Vaccine. 2009 Nov 5;27(47):6589-94. doi: 10.1016/j.vaccine.2009.08.032. Epub 2009 Aug 27. PMID 19716456
- [Derived] Rajendran M, Nachbagauer R, Ermler ME, Bunduc P, Amanat F, Izikson R, Cox M, Palese P, Eichelberger M, Krammer F. Analysis of Anti-Influenza Virus Neuraminidase Antibodies in Children, Adults, and the Elderly by ELISA and Enzyme Inhibition: Evidence for Original Antigenic Sin. mBio. 2017 Mar 21;8(2):e02281-16. doi: 10.1128/mBio.02281-16. PMID 28325769
- [Derived] Nachbagauer R, Choi A, Izikson R, Cox MM, Palese P, Krammer F. Age Dependence and Isotype Specificity of Influenza Virus Hemagglutinin Stalk-Reactive Antibodies in Humans. mBio. 2016 Jan 19;7(1):e01996-15. doi: 10.1128/mBio.01996-15. PMID 26787832
- See also: Related Info — http://proteinsciences.com